CLINICAL TRIAL: NCT03255941
Title: 'A Randomized Controlled Trial of Safety and Effectiveness of Depo Provera Intramuscular and Subcutaneous Administration Comparing Lay Lady Health Workers With Clinically-trained Family Welfare Workers in Pakistan
Brief Title: Clinical Study of Depo Provera Comparing Lay Health Workers and Clinically-trained Health Workers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Aga Khan University (Other); Jhpiego (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Population Welfare Department, Government of Sindh, Pakistan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4798-CHS-ERC-17
Record Dates: First submitted 2017-07-19; First posted 2017-08-21 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Contraception
Keywords: FWW (Family Welfare Worker); LHW (Lady Health Worker); DMPA (Depot medroxyprogesterone acetate or Depo Provera); DMPA IM (Depo Provera intramuscular injection); SP (Sayana Press subcutaneous injection); Contraception; CBA2I (Community-based access to injectables); Sayana (Sayana Press); JHPIEGO (Johns Hopkins Program for International Education in Gynaecology and Obstetrics); Sayana
MeSH Terms: interventions — N,N-dimethyl-4-anisidine

STUDY DESIGN:
Intervention Model Description: Women who are new users of injectable contraception will be randomly assigned to receive services from an LHW or an FWW and will be randomly assigned to receive either intramuscular DMPA or the subcutaneous formulation, Sayana Press.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Clinic Provider - Urban (Active Comparator): Urban Clinic Provider providing DMPA or Sayana Press
  Interventions: Drug: DMPA; Drug: Sayana Press
- Lay Provider - Urban (Active Comparator): Urban Lay Provider providing DMPA or Sayana Press
  Interventions: Drug: DMPA; Drug: Sayana Press
- Clinic Provider- Rural (Active Comparator): Rural Clinic Provider providing DMPA or Sayana Press
  Interventions: Drug: DMPA; Drug: Sayana Press
- Lay Provider- Rural (Active Comparator): Rural Lay Provider providing DMPA or Sayana Press
  Interventions: Drug: DMPA; Drug: Sayana Press

INTERVENTIONS:
Drug: DMPA — The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA.
Drug: Sayana Press — The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press

SUMMARY:
This is a randomized controlled trial comparing lay Lady Health Workers (Lay Health Workers) with Family Welfare Workers (Clinically- trained Health Workers) on quantitative measures of safety and effectiveness of Depo Provera and Sayana Press provision in a clinic setting. This comparative trial will test the non-inferiority hypothesis that Lady Health Workers are just as competent as clinically-trained Family Welfare Workers in screening and counseling first-time injectable users. These first time users will also be randomly assigned to receive intramuscular or subcutaneous injections of DMPA.

DETAILED DESCRIPTION:
FHI 360 and Jhpiego in collaboration with USAID, Aga Khan University (AKU) and the Government of Sindh province propose a randomized controlled trial (RCT) to provide evidence that could change current policies in Pakistan that forbid initiation of DMPA by Lady Health Workers (LHWs). Positive findings on the safety and effectiveness of LHW-initiation of DMPA may also prompt the WHO to consider modifying the recommendation for targeted M&E for lay health worker provision of intramuscular injectable contraceptives. The trial will compare the screening and counseling of (LHWs)-the main lay health worker cadre--with that of Family Welfare Workers (FWWs) who are clinically-trained. The Government of Sindh province also expressed interest in introducing Pfizer's subcutaneous form of Depo Provera, Sayana Press® (SP) in Pakistan, which could simplify administration of injectable contraceptives. As such, an SP arm will be included in the trial, which will be facilitated by relevant training of LHWs and FWWs by Jhpiego and stocks provided by a special USAID procurement, since the registration process for SP in Pakistan is ongoing. A successful RCT demonstrating the non-inferiority of LHWs vis á vis FWWs on first-dose initiation of Depo Provera IM (DMPA IM) and (SP) would facilitate efforts to expand CBA2I in Pakistan, and in turn improve access to family planning services for a potentially large number of underserved women.

ELIGIBILITY:
Inclusion Criteria:

* Women who voluntarily accept DMPA

Exclusion Criteria:

* Women unable to provide informed consent
* Women with contraindications to DMPA
* Women who are pregnant

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Gender at birth
Enrollment: 460 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn S Chin-Quee, PhD, MPH, Principal Investigator — FHI 360
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 461 participants were assessed for eligibility and 460 were randomized to a provider.
Groups:
- Clinic Provider - Urban: Family Welfare Workers that are clinically trained providers in the urban setting of Karachi
- Lay Provider - Urban: Lady Health Workers that are not clinically trained in the urban setting of Karachi
- Clinic Provider - Rural: Famly Welfare Workers that are clinically trained providers in the rural setting of Thatta
- Lay Provider - Rural: Lady Health Workers that are not clinically trained providers in the rural setting of Thatta
Period: Overall Study
Arm/Group | Clinic Provider - Urban | Lay Provider - Urban | Clinic Provider - Rural | Lay Provider - Rural
Started (The 460 randomized participants were equally randomized between lay health workers and clinical providers. These 460 were then assessed by the gold standard nurse and 92 participants were deemed to be not eligible or refused injection.) | 177 | 178 | 53 | 52
Deemed Eligible to Receive DMPA | 140 | 134 | 48 | 46
Completed | 139 | 132 | 48 | 46
Not Completed | 38 | 46 | 5 | 6
Not completed — Not eligible or refused injection | 37 | 44 | 5 | 6
Not completed — Did not complete exit interview | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clinic Provider Urban; Clinic Provider Rural; Lay Provider Rural: Clinic provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA or Sayana Press.
- Lay Provider Urban: Lay Provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA or Sayana Press.
- Total: Total of all reporting groups
Arm/Group | Clinic Provider Urban | Lay Provider Urban | Clinic Provider Rural | Lay Provider Rural | Total
Number analyzed (Participants) | 177 | 178 | 53 | 52 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (5.4) | 27.1 (6.0) | 30.1 (30.1) | 29.7 (5.2) | 28.14 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Only females as participants who accepted intramuscular or subcutaneous DMPA.
  Participants
    Female | 177 | 178 | 53 | 52 | 460
    Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — There were 2 regions in Pakistan: Karachi which is urban and Thatta which is rural.
  participants
    Pakistan | 177 | 178 | 53 | 52 | 460

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Appropriately Screened for Contraceptive Use
Description: Number of participants that were appropriately screened for injectable contraceptive use in both rural and urban settings in Pakistan.
Time Frame: 3 months from randomization
Population: Clients of lay providers or clinic providers who are screened appropriately for injectable contraceptive use
Measure: Count of Participants; unit: Participants
Groups:
- Clinic Provider - Urban: Urban Clinic Provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA or Sayana Press.
- Lay Provider - Urban: Urban Lay Provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press or DMPA
- Clinic Provider - Rural: Rural Clinic Provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press or DMPA
- Lay Provider - Rural: Rural Lay Provider providing DMPA or Sayana Press
  The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press or DMPA
Arm/Group | Clinic Provider - Urban | Lay Provider - Urban | Clinic Provider - Rural | Lay Provider - Rural
Number analyzed (Participants) | 176 | 176 | 52 | 52
Participants
  Screening appropriate | 155 | 136 | 49 | 51
  Screening not appropriate | 21 | 40 | 3 | 1

2. Primary Outcome: Number of Participants That Were Appropriately Counseled for DMPA Use.
Description: Number of participants that were appropriately counseled by both types of providers in both urban and rural settings.
Time Frame: 3 months from randomization
Population: Clients of lay and clinic providers who receive appropriate counseling for Injectable contraceptive use.
Measure: Count of Participants; unit: Participants
Groups:
- Clinic Providers - Urban: Appropriateness of counseling by Urban Clinic providers.
- Lay Provider - Urban: Appropriateness of counseling by Urban Lay providers.
- Clinic Provider - Rural: Appropriateness of counseling by Rural Clinical Providers
- Lay Provider - Rural: Appropriateness of counseling by Rural Lay Providers
Arm/Group | Clinic Providers - Urban | Lay Provider - Urban | Clinic Provider - Rural | Lay Provider - Rural
Number analyzed (Participants) | 177 | 178 | 53 | 52
Participants
  Counseling appropriate | 17 | 24 | 24 | 29
  Counseling not appropriate | 160 | 154 | 29 | 23

3. Secondary Outcome: Proportion of Clients Providers Who Report Satisfaction With the DMPA Method Received From the Provider
Description: DMPA clients served by both types of providers in both urban and rural settings will report whether or not they were satisfied with the DMPA method provided to them.
Time Frame: 3 months from randomization
Population: Clients of lay and clinic providers reports of satisfaction with the DMPA method received.
Measure: Count of Participants; unit: Participants
Groups:
- DMPA - IM Urban; DMPA-IM Rural: Provider providing DMPA- Intra muscular
  Proportion of clients highly satisfied with their DMPA Method
- DMPA - SC - Urban; DMPA-SC- Rural: Provider providing DMPA - sub cutaneous
  Prop[portion of clients highly satisfied with the DMPA method provided to them
Arm/Group | DMPA - IM Urban | DMPA - SC - Urban | DMPA-IM Rural | DMPA-SC- Rural
Number analyzed (Participants) | 135 | 139 | 45 | 49
Participants | 107 | 108 | 41 | 42

4. Secondary Outcome: Proportion of Clients Who Report Satisfaction With Provider Services
Description: Clients who received intramuscular or subcutaneous DMPA injections will report whether or not they were satisfied with the services provided to them by their provider.
Time Frame: 3 months from randomization
Population: Clients of lay and clinic providers who report satisfaction with DMPA services provided by their provider.
Measure: Count of Participants; unit: Participants
Groups:
- Clinic Provider - Urban: Urban Clinic provider providing DMPA services
- Lay Provider- Urban: Urban Lay provider providing DMPA services
- Clinic Provider - Rural: Rural Clinic provider providing DMPA services
- Lay Provider - Rural: Lay rural provider providing DMPA services
Arm/Group | Clinic Provider - Urban | Lay Provider- Urban | Clinic Provider - Rural | Lay Provider - Rural
Number analyzed (Participants) | 139 | 132 | 48 | 46
Participants | 125 | 112 | 42 | 40

ADVERSE EVENTS:
Time Frame: This study was cross-sectional; no adverse events data were collected.
Groups:
- Lay Provider & DMPA: Lay provider providing DMPA
  DMPA: The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA.
- Lay Provider & Sayana Press: Lay Provider providing Sayana Press
  Sayana Press: The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press
- Clinic Provider & DMPA: Clinic provider providing DMPA
  DMPA: The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use DMPA.
- Clinic Provider and Sayana Press: Clinic provider providing Sayana Press
  Sayana Press: The safety and effectiveness of provision of injectable contraception will be compared between providers' screening and counseling for eligibility to use Sayana Press
Arm/Group | Lay Provider & DMPA | Lay Provider & Sayana Press | Clinic Provider & DMPA | Clinic Provider and Sayana Press
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03255941/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT03255941/SAP_001.pdf